CLINICAL TRIAL: NCT04634747
Title: A Single-Arm, Open-Label, Multi-Center Phase II Study to Evaluate the Combination of PVX-410 + Pembrolizumab + Chemotherapy for Frontline Therapy of Metastatic, PD-L1+ Triple-Negative Breast Cancer (TNBC) in HLA-A2-Positive Patients
Brief Title: Phase 2 Study to Evaluate PVX-410 + Pembrolizumab + Chemotherapy for Metastatic, PD-L1+ Triple-Negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: OncoPep, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-001
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — PVX-410 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PVX-410/pembrolizumab/chemotherapy (Experimental)
  Interventions: Drug: PVX-410

INTERVENTIONS:
Drug: PVX-410 — PVX-410 in combination with pembrolizumab and chemotherapy

SUMMARY:
Evaluating the combination of the investigational, multi-peptide cancer vaccine PVX-410 in combination with pembrolizumab and chemotherapy in treatment naive patients with metastatic, triple negative breast cancer who are PDL1 and HLA A2 positive.

ELIGIBILITY:
Inclusion Criteria:

- HLA A2 Positive PDL1 Positive Treatment naive, triple negative breast cancer

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2022-04-30 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 8 months

IPD SHARING:
Plan to Share IPD: No